CLINICAL TRIAL: NCT01632176
Title: A Brief Intervention to Prevent Adolescent Dating Aggression Perpetration
Brief Title: A Brief Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5K01AA017630-04 (NIH); K01AA017630 (NIH)
Record Dates: First submitted 2012-06-28; First posted 2012-07-02 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Dating Violence; Dating Abuse
Keywords: dating abuse; dating violence; domestic violence; sexual violence; sexual assault; youth violence; underage alcohol use; alcohol use
MeSH Terms: conditions — Underage Drinking; Alcohol Drinking | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): Patients in the control group will not receive any intervention, but will receive standard care for dating abuse issues.
- Intervention (Experimental): Patients in the intervention group will participate in brief, motivational interview and one booster session to prevent adolescent dating abuse.
  Interventions: Behavioral: Brief, motivational interview and one booster session

INTERVENTIONS:
Behavioral: Brief, motivational interview and one booster session — This is a one session brief motivational interview-style intervention that follows a 9-step intervention algorithm. The intervention is delivered by a trained motivational interview interventionist. There is one booster call 10 days after the intervention/
  Arms: Intervention

SUMMARY:
This randomized controlled trial (RCT) study is a small scale test of the feasibility and preliminary efficacy of a brief motivational interview-style intervention. The intervention took place in the pediatric emergency departments by a trained interventionist and will followed an intervention algorithm developed by a team of dating abuse and brief intervention experts. The research design is as follows: the investigators will randomize youth ages 12-19 years old to one of two groups: one group who receives the intervention (N=~18), and the other which does not (N=~18). The investigators compared changes in outcomes from baseline to 1-month follow-up for those in both groups. The investigators looked at outcomes including dating abuse-related knowledge, attitudes about the use of violence to resolve conflict, and dating abuse behavior (perpetration and/or victimization).

Statement of study hypothesis: Youth who receive the intervention will show improvements in dating abuse-related knowledge, attitudes and behavior that are maintained for 1 month, while those in the comparison group will show no similar change.

ELIGIBILITY:
Inclusion Criteria:

* 15-19 years old
* English-speaking
* Have used at least one form of physical or sexual aggression against a dating or sexual partner in the past three months

Exclusion Criteria:

* Patient's reason for ED visit is an acute mental health problem (e.g., suicidal ideation or attempt, severe anxiety attack)
* Patient is a prisoner
* Patient is determined to be potentially lethal
* Patient attends batterer intervention classes

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2013-01 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Dating abuse perpetration | 1 month
  Self-reported perpetration of dating abuse, including acts such as pushing, hitting, kicking and forcing partner to have sex.

CONTACTS AND LOCATIONS:
Overall Officials: Emily F Rothman, ScD, Principal Investigator — Boston University
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rothman EF, Wang N. A feasibility test of a brief motivational interview intervention to reduce dating abuse perpetration in a hospital setting. Psychol Violence. 2016 Jul;6(3):433-441. doi: 10.1037/vio0000050. Epub 2016 Mar 24. PMID 27525169